CLINICAL TRIAL: NCT07145723
Title: Supporting Care Partners' Well-Being With AI Chatbots: A Feasibility and Acceptability Study
Brief Title: Supporting Care Partners' Well-Being With Artificial Intelligence (AI) Chatbots
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Mark Newman, Professor of Information, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00271412
Record Dates: First submitted 2025-08-20; First posted 2025-08-28 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Caregivers
Keywords: Caregivers for adults with dementia; Surveys; Care partners; Artificial intelligence (AI) mobile application; Quality of life; Chatbot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Earkick app (Experimental)
  Interventions: Other: Earkick app

INTERVENTIONS:
Other: Earkick app — Participants will have a baseline visit followed by an 8-week home monitoring period (HMP) using the Earkick app.
  The Earkick app will interact with a mental health chatbot. Participants will complete online surveys at the midpoint (4 weeks) and end (8 weeks) of the HMP. Participants will choose one mental health-related topic to focus on from weeks 1-4 and one physical health-related topic to focus on from weeks 5-8.
  Additionally, participants will have a post-HMP interview over Zoom.

SUMMARY:
This study is being completed to test an AI therapy chatbot application called Earkick to see whether it is feasible and acceptable in supporting care partners who support individuals living with dementia.

ELIGIBILITY:
Inclusion Criteria:

* Participants need to be a care partner (informal caregiver) of an individual living with dementia
* Participant provides emotional, physical, and/or financial support/assistance to the individual with dementia (per protocol)
* Participants indicate high levels of caregiver burden, confirmed using the 12-item Zarit Burden questionnaire (per protocol)
* Provide informed consent and read, speak, and understand English
* Have an Apple smartphone, tablet, or laptop, have access to the internet and text messages, and be willing to use this device as well as internet and text message access for the study, including downloading the AI chatbot app
* Be willing to complete all study assessments

Exclusion Criteria:

* Professional, paid caregivers
* Anything that would preclude safe or meaningful participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility and Acceptability as measured by the Feasibility and Acceptability Questionnaire | 4 weeks and 8 weeks (post intervention)
  Feasibility and Acceptability Questionnaire (items are scaled from 1 to 5 to indicate level of agreement, where "1" indicates "strong disagreement" and "5" indicates "strong agreement").

SECONDARY OUTCOMES:
Attrition as measured by the percent of participants completing the study | 8 weeks
Adherence as measured by the percentage of missing data over the course of the study | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Newman, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No